CLINICAL TRIAL: NCT05765851
Title: A Phase 1, 2-Part, Multicenter, First-In-Human Dose-Escalation and Dose-Expansion Study of DS-1103a Combination Therapy in Subjects With Advanced Solid Tumors
Brief Title: A Study of DS-1103a Combination Therapy in Participants With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS1103-074; 2023-503965-48-00 (Other: EU CT)
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor; Breast Cancer
Keywords: Advanced Solid Tumor; Breast Cancer; DS-1103a; CD47; SIRPa
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation: DS-1103a + T-DXd (Experimental): Participants with HER2-expressing or HER2-mutant advanced metastatic solid tumors who will receive an intravenous (IV) infusion of DS-1103a (starting dose of 100 mg) every 3 weeks (Q3W) starting on Cycle 1 Day 1. Starting on Cycle 2 Day 1 and on Day 1 of each subsequent cycle, participants will also receive T-DXd Q3W at a dose of 5.4 mg/kg.
  Interventions: Drug: DS-1103a; Drug: T-DXd
- Dose Expansion: DS-1103a + T-DXd (Experimental): Participants with HER2-low expressing breast cancer who will receive an IV infusion of DS-1103a at the recommended dose for expansion (RDE) in combination with T-DXd 5.4 mg/kg Q3W starting on Cycle 1 Day 1.
  Interventions: Drug: DS-1103a; Drug: T-DXd

INTERVENTIONS:
Drug: DS-1103a — One IV infusion Q3W on Day 1 of each 21-day cycle
Drug: T-DXd — One IV infusion Q3W on Day 1 of each 21-day cycle
  Other Names: DS-8201a (trastuzumab derextecan); Enhertu®

SUMMARY:
This study will evaluate the safety and efficacy of DS-1103a combination therapy in patients with advanced solid tumors.

DETAILED DESCRIPTION:
DS-1103a, a recombinant humanized IgG4 anti-SIRPα antibody designed to block the SIRPα-CD47 interaction, is being developed for the treatment of advanced cancers in combination with other anticancer therapies. This is the first-in-human, dose-escalating clinical study designed to assess the safety and efficacy of DS-1103a combination therapy in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Sign and date the informed consent form (ICF), prior to the start of any study-specific qualification procedures
* Adults ≥18 years of age at the time the ICF is signed (please follow local regulatory requirements if the legal age of consent for study participation is >18 years old)
* Pathologically documented HER2-expressing (immunohistochemistry [IHC] 1+ or greater) or HER2-mutated (activating mutation) solid tumor that is unresectable or metastatic (further detailed in inclusion criteria specific for Part 1 and Part 2 below)
* Is willing and able to provide adequate baseline tumor samples. If an adequate archival tumor tissue is not available, a fresh tumor tissue biopsy is required
* Presence of at least 1 measurable lesion based on computed tomography (CT) or magnetic resonance imaging (MRI) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) by investigator assessment
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Has a left ventricular ejection fraction (LVEF) ≥50% by either an echocardiogram (ECHO) or multigated acquisition (MUGA) scan within 28 days before enrollment
* Has adequate organ and bone marrow function within 28 days before the start of study treatment. Transfusion (red blood cell or platelet) or granulocyte-colony stimulating factor (G-CSF) administration is not allowed within 14 days prior to the start of study treatment.
* If the participant is a female of childbearing potential, she must have a negative serum pregnancy test at Screening and must be willing to use highly effective birth control upon enrollment, during the Treatment Period, and for at least 10 months following the last dose of study drug(s).
* If male, the participant must be surgically sterile or their female partner of childbearing potential must be willing to use highly effective birth control upon enrollment, during the Treatment Period, and for 6 months following the last dose of study drug(s). In addition to the above, it is recommended that the male participant uses a condom throughout this period to prevent their partner from possibly being exposed to the study drug(s) via sperm.
* Male participants must not freeze or donate sperm from the time of enrollment, during the Treatment Period, and for at least 6 months after the final study drug(s) administration
* Female participants must not donate, or retrieve for their own use, ova from the time of enrollment, during the Treatment Period, and for at least 10 months after the final study drug(s) administration
* Is willing and able to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions

Dose-escalation Phase:

* Has progressed or was non-responsive to available therapies and for which no standard or available anticancer therapy exists
* Has a pathologically documented HER2-expressing (eg, breast cancer) or HER2-mutated (eg, non-small cell lung cancer [NSCLC]) solid tumor (participants with gastric cancer or gastroesophageal junction adenocarcinoma are not eligible)

Dose-expansion Phase:

* Pathologically documented breast cancer that:

  * Has a history of low HER2 expression, defined as IHC 2+/in situ hybridization negative (ISH-) or IHC 1+ (ISH- or untested) according to American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) 2018 HER2 testing guidelines
  * Is hormone receptor (HR)-positive or HR-negative (HR-positive for estrogen receptor or progesterone receptor if finding of ≥1% of tumor cell nuclei are immunoreactive), as defined by ASCO/CAP HR testing guidelines
  * Has been treated with at least 1 and at most 2 prior lines of chemotherapy in the recurrent or metastatic setting. If recurrence occurred within 6 months of (neo)adjuvant chemotherapy, (neo)adjuvant therapy would count as 1 line of chemotherapy
  * Was never previously HER2-positive (IHC 3+ or IHC 2+/ISH+) on prior pathology testing (per ASCO/CAP guidelines) or was historically HER2 IHC 0 only
  * Was never previously treated with anti-HER2 therapy
  * Documented radiologic progression (during or after most recent treatment)

Exclusion Criteria:

* Has had prior treatment with an anti-CD47 or anti-signal regulatory protein α (SIRPα) therapy.
* Has an inadequate treatment washout period prior to start of study treatment, defined as follows:

  * Major surgery: ≤4 weeks or ≤2 weeks for low-invasive cases (eg, colostomy)
  * Radiation therapy including palliative stereotactic radiation to chest: ≤4 weeks
  * Palliative stereotactic radiation therapy to other anatomic areas: ≤2 weeks
* Received any systemic agent from a previous treatment regimen or clinical study within the specified time frame prior to administration of study treatment as specified in the protocol
* Medical history of myocardial infarction (MI) within 6 months before study enrollment, symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] Class II to IV
* Has a QT interval corrected with Fridericia's formula (QTcF) prolongation to >470 ms (females) or >450 ms (males) based on average of the screening triplicate 12-lead electrocardiogram (ECG)
* Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening
* Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms
* Has multiple primary malignancies within 3 years, except adequately resected non-melanoma skin cancer, curatively treated in-situ disease, other solid tumors curatively treated, or contralateral breast cancer
* Has a history of severe hypersensitivity reactions to either the drug substances or inactive ingredients in the drug products or other monoclonal antibodies
* Has an uncontrolled infection requiring intravenous (IV) antibiotics, antivirals, or antifungals
* Is requiring concomitant use of chronic systemic (IV or oral) corticosteroids or other immunosuppressive medications during the study
* Has received a live, attenuated vaccine (messenger ribonucleic acid [mRNA] and replication-deficient adenoviral vaccines are not considered live, attenuated vaccines) within 30 days prior to first exposure to study drug(s)
* Has substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the participant's participation in the clinical study or evaluation of the clinical study results.
* Has active primary immunodeficiency or active human immunodeficiency virus (HIV) infection as determined by plasma HIV ribonucleic acid (RNA) viral load and CD4 count. For the Dose-expansion phase only, participants with undetectable viral load or normalized CD4 count (CD4+ T-cell counts ≥ 350 cells/μL) and no opportunistic infection within the past 12 months will be eligible. These participants must be on established antiretroviral therapy for at least 4 weeks and have an HIV viral load <400 copies/mL prior to enrollment.
* Has active hepatitis B or C infection. Participants with past hepatitis C virus (HCV) infection and positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA. Participants with past or resolved hepatitis B virus infection are eligible only if they meet pre-specified criteria.
* Has unresolved toxicities from previous anticancer therapy
* Female who is pregnant, breastfeeding, or planning to become pregnant
* Has lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder
* Any autoimmune, connective tissue or inflammatory disorders where there is documented or a suspicion of pulmonary involvement at the time of Screening
* Prior complete pneumonectomy
* Any of the following within 6 months of enrollment: Cerebrovascular accident, transient ischemic attack, other arterial thromboembolic event, or pulmonary embolism
* Psychological, social, familial, or geographical factors that would prevent regular follow-up
* Any active or chronic corneal disorders, other active ocular conditions requiring ongoing therapy, or any clinically significant corneal disease that prevents adequate monitoring of drug-induced keratopathy
* Uncontrolled hypertension (resting systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg) and/or severe arrhythmia within 28 days before enrollment

Dose-escalation Phase:

* Same as noted above for overall study

Dose-expansion Phase:

* Has had prior treatment with antibody-drug conjugate that consists of an exatecan derivative that is a topoisomerase I inhibitor including prior participation in a study involving an antibody-drug conjugate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicities Following DS-1103a Combination Therapy (Dose Escalation) | From Cycle 1 Day 1 up to 3-month safety follow up (each cycle is 21 days)
Overall Number of Participants With Treatment-emergent Adverse Events and Serious Adverse Events Following DS-1103a Combination Therapy (Dose Expansion) | Screening (Day -28 to 0) through long-term follow up, up to approximately 44 months
Number of Participants With Objective Response Rate Assessed by Blinded Independent Central Review Following DS-1103a Combination Therapy (Dose Expansion) | Baseline up until documented progressive disease, unacceptable toxicity, death, lost to follow-up, or withdrawal by the participant, up to approximately 44 months
  Confirmed objective response rate (ORR) is defined as the sum of the complete response (CR) rate and partial response (PR) rate based on blinded independent central review (BICR) by Response Evaluation Criteria In Solid Tumors v1.1 and confirmed by a second assessment.

SECONDARY OUTCOMES:
Number of Participants With Objective Response Rate Assessed by Investigator Following DS-1103a Combination Therapy (Dose Escalation and Dose Expansion) | Baseline up until documented progressive disease, unacceptable toxicity, death, lost to follow-up, or withdrawal by the participant, up to approximately 44 months
  Confirmed objective response rate (ORR) is defined as the sum of the complete response (CR) rate and partial response (PR) rate based on investigator (Response Evaluation Criteria In Solid Tumors v1.1) and confirmed by a second assessment.
Disease Control Rate Following DS-1103a Combination Therapy Assessed by Investigator (Dose Escalation) or Blinded Independent Central Review (Dose Expansion) | Baseline up until documented progressive disease, unacceptable toxicity, death, lost to follow-up, or withdrawal by the participant, up to approximately 44 months
  Disease control rate is defined as the sum of the CR rate, PR rate, and stable disease (SD) rate based on investigator assessment (Dose Escalation) or blinded independent central review (BICR)(Dose Expansion).
Clinical Benefit Rate Following DS-1103a Combination Therapy (Dose Escalation and Dose Expansion) | Baseline up until documented progressive disease, unacceptable toxicity, death, lost to follow-up, or withdrawal by the participant, up to approximately 44 months
  Clinical benefit rate (CBR) is defined as the sum of the CR rate, PR rate, and ≥6 months SD rate based on investigator assessment (Dose Escalation) or BICR (Dose Expansion).
Duration of Response Following DS-1103a Combination Therapy (Dose Escalation and Dose Expansion) | Baseline up until documented progressive disease, unacceptable toxicity, death, lost to follow-up, or withdrawal by the participant, up to approximately 44 months
  Duration of response (DoR) is defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first documentation of progressive disease (PD) (based on investigator assessment [Dose Escalation] or blinded independent central review (BICR) [Dose Expansion]) or death. The DoR will be calculated for responding participants (PR or CR) only.
Pharmacokinetic Parameter Area Under the Plasma Concentration Curve for DS-1103a (Dose Escalation and Dose Expansion) | Dose Escalation: Cycles 1,2, and 4: Days 1,2,4,8,15; Cycle 3 Days 1,8,15; Cycle 5 and beyond Day 1; Dose Expansion: Cycles 1 and 3: Days 1,2,4,8,15; Cycle 2 Days 1,8,15; Cycle 4 and beyond Day 1 (each cycle is 21 days)
  Area under the plasma concentration-time curve up to the last quantifiable time (AUClast) and Area under the plasma concentration-time curve during dosing interval (AUCtau) will be assessed using non-compartmental methods.
Pharmacokinetic Parameter Maximum Plasma Concentration for DS-1103a (Dose Escalation and Dose Expansion) | Dose Escalation: Cycles 1,2, and 4: Days 1,2,4,8,15; Cycle 3 Days 1,8,15; Cycle 5 and beyond Day 1; Dose Expansion: Cycles 1 and 3: Days 1,2,4,8,15; Cycle 2 Days 1,8,15; Cycle 4 and beyond Day 1 (each cycle is 21 days)
  Maximum plasma concentration (Cmax) will be assessed using non-compartmental methods.
Pharmacokinetic Parameter Time to Maximum Plasma Concentration for DS-1103a (Dose Escalation and Dose Expansion) | Dose Escalation: Cycles 1,2, and 4: Days 1,2,4,8,15; Cycle 3 Days 1,8,15; Cycle 5 and beyond Day 1; Dose Expansion: Cycles 1 and 3: Days 1,2,4,8,15; Cycle 2 Days 1,8,15; Cycle 4 and beyond Day 1 (each cycle is 21 days)
  Time to maximum plasma concentration (Tmax) will be assessed using non-compartmental methods.
Pharmacokinetic Parameter Minimum Plasma Concentration for DS-1103a (Dose Escalation and Dose Expansion) | Dose Escalation: Cycles 1,2, and 4: Days 1,2,4,8,15; Cycle 3 Days 1,8,15; Cycle 5 and beyond Day 1; Dose Expansion: Cycles 1 and 3: Days 1,2,4,8,15; Cycle 2 Days 1,8,15; Cycle 4 and beyond Day 1 (each cycle is 21 days)
  Minimum plasma concentration (Cmin) will be assessed using non-compartmental methods.
Number of Participants With Treatment-emergent Anti-drug Antibodies Following DS-1103a Combination Therapy (Dose Escalation and Dose Expansion) | Predose on Cycles 1 to 2 (Days 1, 15), Cycles 3 and 4 (Day 1), thereafter every 2 cycles (Day 1), end of treatment, 40-day safety follow-up, and every 3 months, up to 1 year from last dose or until anti-drug antibodies are negative (each cycle, 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (8):
- United States (4):
  - Florida Cancer Specialists, Sarasota, Florida
  - Lifespan Cancer Institute, Providence, Rhode Island
  - University of Utah, Salt Lake City, Utah
  - NEXT Oncology, Fairfax, Virginia
- Princess Margaret Cancer Centre, University Health Network, Toronto, Canada
- France (2):
  - Oncopole - Institut Claudius Regaud, Toulouse, Haute Garonne
  - Centre Léon Bérard, Lyon, Rhone
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/